CLINICAL TRIAL: NCT04223037
Title: Phase III Clinical Trial of Purified Inactivated Japanese Encephalitis Vaccine
Brief Title: Purified Inactivated Japanese Encephalitis Vaccine
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mingbo Sun, Director， WHO Prequalification Department, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 074201504
Record Dates: First submitted 2020-01-06; First posted 2020-01-10 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Japanese Encephalitis Virus Disease
Keywords: Japanese Encephalitis Vaccine; Phase III Clinical Trial
MeSH Terms: conditions — Encephalitis, Japanese | interventions — Japanese Encephalitis Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Day 0，7 immunization shedule (Active Comparator): Japanese Encephalitis Vaccine produced by Institute of Medical Biology, Chinese Academy of Medical Sciences (IMBCAMS) and Japanese Encephalitis Vaccine produced by Liaoning Chenda CO.,LTD Dosage form: 0.5mL/vial Two Dose injection with 7 days interval
  Interventions: Biological: Japanese Encephalitis Vaccine produced by IMBCAMS; Biological: Japanese Encephalitis Vaccine produced by Liaoning Chenda
- Day 0，28 immunization shedule (Experimental): Japanese Encephalitis Vaccine produced by IMBCAMS Dosage form: 0.5mL/vial Two Dose injection with 28 days interval
  Interventions: Biological: Japanese Encephalitis Vaccine produced by IMBCAMS

INTERVENTIONS:
Biological: Japanese Encephalitis Vaccine produced by IMBCAMS — Dosage form: 0.5mL/vial
Biological: Japanese Encephalitis Vaccine produced by Liaoning Chenda — Dosage form: 0.5mL/vial
  Arms: Day 0，7 immunization shedule

SUMMARY:
This study evaluates the immunogenicity and safety of a purified inactivated JE vaccine compared to a commercialized JE vaccine. In this phase III, randomized, blind trial, infants at 6-23 months of age were randomly assigned to three groups to receive experimental vaccine or control vaccine with two different vaccination schedule respectively.

DETAILED DESCRIPTION:
The clinical study used randomized, blind method, commercialize inactivated Japanese encephalitis vaccine as control. In Infants at 6-23 months of age were injected with experimental vaccine with 0,7 days and 0,28 days vaccination schedule to evaluate immunogenicity and safety of the experimental vaccine and the effectiveness of different vaccination schedule. Participates were assigned to three groups (350 per group): group 1 with experimental vaccine using 0,7 days vaccination schedule; group 2 with control vaccine using 0, 7 days vaccination schedule; group 3 with experimental vaccine using 0, 28 vaccination schedule.

Blood samples were collected before immunization and 30 days after immunization, and the neutralization antibody of Japanese encephalitis was detected by plaque reduction neutralization test. Medical observation was conducted 30 minutes after each injection. Body temperature of participates was continuously measured for 7 days, and any adverse events were observed and recorded from the first dose to 30 days after the whole vaccination. Serious adverse events were collected within 6 months after the first dose.

ELIGIBILITY:
Inclusion Criteria:

* 6-23 months old infants, no vaccination history of JE vaccine, no vaccination contraindication.
* informed consent of guardian / lawful written guardian, and signed informed consent;
* the guardian and family can comply with the requirements of the clinical trial scheme.
* there was no immunization history of immunoglobulins within three months, and there was no history of live vaccination within 14 days.
* the axillary temperature ≤ 37℃.

Exclusion Criteria:

* Allergy to any ingredient in the vaccine (any previous history of vaccine allergy); There are allergic, convulsive, epileptic, encephalopathy and psychiatric symptoms or signs.
* People with known or suspected (or high-risk) impairment or abnormality of immune function, such as those receiving immunosuppressive or immunopotentiator therapy, receiving blood products or plasma extracts within three months, or having an immunodeficiency virus infection or related disease in the mother or child.
* A history of thrombocytopenia or other coagulation disorders clearly diagnosed by the medical department, or a history of hemorrhagic constitution or prolonged bleeding time;
* Infected patients with known or suspected to have respiratory diseases, acute infections or active chronic diseases and are receiving antibiotic or antiviral treatment;
* In the past 3 days, fever (axillary body temperature≥38℃), oral or steroid hormones were given.
* Infectious or allergic skin diseases.
* Participating in another clinical researcher; or any situation that the researcher considers likely to affect the evaluation of the trial

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1050 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Local and systemic adverse reactions | Within 6 months after immunization
  The main endpoint of safety observation was 30 days after 2 doses vaccination. If serious adverse reactions related to vaccines occur during the observation period, or the adverse reactions of grade 3 and above reached 10%, or three symptoms similar to grade 3 and above occur within 24 hours, the trial should be suspended and vaccine-related adverse reactions occurred. The death of the subjects will be terminated at any time. Follow up and collection of serious adverse events within 6 months after first dose immunization via close monitoring or diary card.
Immunogenecity detected by plaque reduction neutralization test | 1 month after immunization
  Blood samples were collected from all subjects before and 30 days after the whole course of immunization, and neutralizing antibody was detected by plaque reduction neutralization test.

CONTACTS AND LOCATIONS:
Overall Officials: Shaohong Yan, Principal Investigator — Disease prevention and control center of Inner Mongolia autonomous region
Locations (1):
- Disease prevention and control center of Inner Mongolia autonomous region, Hohhot, Inner Mongolia, China